CLINICAL TRIAL: NCT03292744
Title: Effect of Alfacalcidol Supplementation to Respiratory Infection, Inflammatory Markers and CD4/CD8 Ratio of Indonesian Elderly
Brief Title: Effect of Alfacalcidol to Respiratory Infection and Immune Response of Indonesian Elderly
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aulia Rizka, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VitaminDIndonesia
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Frail Elderly Syndrome; Elderly Infection
Keywords: immunosenescence
MeSH Terms: interventions — alfacalcidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alfacalcidol (Experimental): Alfacalcidol 0,5 mcg once daily for 90 days
  Interventions: Drug: Alfacalcidol
- Placebo (Placebo Comparator): Amylum same capsule form, weight and colour with treatment arm
  Interventions: Drug: Alfacalcidol

INTERVENTIONS:
Drug: Alfacalcidol — alfacalcidol 0,5 mcg
  Other Names: 1 alpha hydroxy cholecalciferol

SUMMARY:
Vitamin D has been known to influence immune response through Vitamin D Receptor in Immune Cells, but only few has been known about the effect alfacalcidol, a vitamin D analog to immune system. In elderly, immune disregulation or immunosenecence have great impact to infection response. This study is aimed to determine the effect of alfacalcidol supplementation in vitro and in vivo to respiratory infection incidence and inflammatory markers, as well as T cell lymphocyte subset in Indonesian elderly patients.

DETAILED DESCRIPTION:
This study consist of 2 designs. First is in vitro study to investigate the effect of alfacalcidol supplementation to IL-6, IL-10 and IFN gamma regulation in Peripheral Blood Mononuclear Cells (PBMC) of elderly and second design is randomised controlled trial to evaluate the effect of 3 months supplementation of alfacalcidol 0,5 mcg in respiratory infection, antibiotic use, inflammatory markers, CD4/CD8 ratio and CD8+ CD28+ in Indonesian elderly with various level of frailty syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Elderly age more than 60
* Willing to join research

Exclusion Criteria:

* In acute infection
* Using NSAID or steroid
* Liver failure
* Hypercalcemia

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-10-10 (Estimated); Study Completion 2017-12-15 (Estimated)

PRIMARY OUTCOMES:
upper respiratory tract infection incidence | 90 days
  incidence of URTI
lower respiratory tract infection incidence | 90 days
  incidence of LRTI

SECONDARY OUTCOMES:
inflammatory markers | day 90
  IL6, IL10 and IFN gamma in PBMC
T cell subset | day 90
  CD4/CD8 ratio, CD8+ CD28- percentage
antibiotic use | 90 days
  any antibiotic prescribed by physician

CONTACTS AND LOCATIONS:
Overall Officials: Aulia Rizka, MD, Principal Investigator — Universitas Indonesia / Cipto Mangunkusumo Hospital
Locations (1):
- Cipto Mangunkusumo National Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No